CLINICAL TRIAL: NCT04244305
Title: Endurance Training in Patients Undergoing Lung Transplantation: Differences Between Treadmill and Cycle Ergometry Training
Brief Title: Endurance Training in Patients Undergoing Lung Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital A Coruña (Other)
Responsible Party: Principal Investigator, Esther Gimenez Moolhuyzen, Principal Investigator, University Hospital A Coruña
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EGM-TXP-2016
Record Dates: First submitted 2019-12-27; First posted 2020-01-28 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Lung Transplantation
Keywords: Exercise Therapy; Physical Therapy Modalities; Functional Capacity
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors were blinded to group allocation of the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill Training (Experimental): Participants in the treadmill training group will perform endurance training during the post-operative period using a treadmill (Salter Housewares, UK) for a minimum of 20 sessions. Intensity of training will be set according to 80% of the mean speed achieved during the 6MWT for a targeted time of 30 minutes. Intensity and duration will be adapted to the participant's physical condition, especially during the first week.
  After the endurance training, participants will perform resistance training for 20 - 30 minutes for conditioning of the main muscles in the upper and lower limbs using elastic bands, dumbbells and body-weight exercises. Intensity will progressively increase up to 70% of the maximum isometric strength measured with a hand-held dynamometer. Volume of training will also increase from 1 to 3 sets of 12 repetitions each. When needed patients will also be taught breathing exercises and airway clearance techniques.
  Interventions: Other: Exercise Therapy
- Cyclo-ergometry Training (Active Comparator): Participants in this group will perfom endurance training during the post-operative period using a cycle ergometer (Monark 828e, Monark AB, Sweeden) for a minimum of 20 sessions. Intensity of training will be set according to the results of a symptom-limited incremental cycle-ergometry test performed on the first day to achieve 80% of the maximal workload obtained for a targeted time of 30 minutes. Intensity and duration will be adapted to the participant's physical condition, especially during the first week. Participants in this group will also perfom resistance training and breathing exercises as in the treadmill training group.
  Interventions: Other: Exercise Therapy

INTERVENTIONS:
Other: Exercise Therapy — Endurance training in the form of treadmill/cycle-ergometry

SUMMARY:
Lung Transplantation is usually the last option for patients with chronic respiratory conditions in the late stages of the disease. Pulmonary rehabilitation and, particularly, endurance training, is a cornerstone in the management of these patients both during the pre-operative as well as the post-operative period as it improves cardiopulmonary fitness, muscle mass, muscle strength, health-related quality of life and potentially, survival. However, very few studies have been published addressing which modality of training, intensity, frequency or duration of training provides the best possible results in these patients. Therefore, the objective of this study was to compare two training modalities (treadmill walking versus cycle-ergometry) on functional capacity, muscle strength and lung function.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lung transplantation at the Thoracic Surgery Unit of the Hospital Clínico Universitario de A Coruña.
* Adults > 18 years.
* Ability to attend post-surgery exercise training for a minimum period of one month.
* Sign informed consent.

Exclusion Criteria:

* Torpid post-operative recovery with a prolonged stay at the Post-Anaesthesia Care Unit > 12 days.
* Diagnosed with intensive care unit acquired muscle weakness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walk Test | 1 month
  Distance covered during the 6 Minute Walk Test performed according to the American Thoracic Guidelines.

SECONDARY OUTCOMES:
6 Minute Walk Test | 3 Months
  Distance covered with the 6 Minute Walk Test performed according to the American Thoracic Guidelines.
Maximal isometric strength | 1 and 3 months
  Isometrical maximal strength of the brachial biceps and quadriceps muscle of both dominant and non-dominant limbs. Maximal isometric strength will be assessed using a hand-held dynamometer (Lafayette Instrument, Model 01165) and will be presented in kilograms
Sit-to-stand | 1 and 3 months
  Number of times the patient can stand up from a chair and sit back in 30 seconds
Forced Expiratory Volume 1st second (FEV1) | 1 and 3 months
  Changes in Forced Expiratory Volume in the 1st second assessed during a forced spirometry test performed according to the international guidelines.
Incremental Symptom-Limited Test | 1 and 3 months
  Incremental symptom-limited test performed on a cycle-ergometry with a 5-10W increase per minute up to maximal tolerance. Patient was monitorised during the test for both heart rate and oxygen saturation.
Maximal inspiratory and expiratory pressures | 1 and 3 months
  Maximal inspiratory and expiratory pressures performed with the respiratory muscles
Forced Expiratory Capacity (FVC) | 1 and 3 months
  Changes in forced expiratory capacity assessed during a forced spirometry test performed according to the international guidelines.
Peak Expiratory Flow (PEF) | 1 and 3 months
  Changes in peak expiratory flow assessed during a forced spirometry test performed according to the international guidelines.

IPD SHARING:
Plan to Share IPD: No